CLINICAL TRIAL: NCT05181722
Title: Evaluating the Use of Patient Navigation to Promote Timely Diagnostic Evaluation During the COVID-19 Pandemic
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Association of University Radiologists (AUR) - GERRAF (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: IRB00313835
Record Dates: First submitted 2022-01-04; First posted 2022-01-06 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Study participants will be randomly assigned to either the usual care group or the intervention group.
Who Masked: Care Provider, Investigator
Masking Description: The patient navigator and statistician will be unblinded to the patient groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): The study participants in this group will receive support from the patient navigator as part of this study.
  Interventions: Other: Patient navigator support
- Usual care group (No Intervention): The study participants in this group will receive the usual care per the institutional protocol.

INTERVENTIONS:
Other: Patient navigator support — Support of a patient navigator for patients who have experienced an abnormal screening mammogram
  Arms: Intervention group

SUMMARY:
The primary objective of this project is to evaluate the role of patient navigation in promoting timely follow-up of abnormal breast imaging findings in patient populations that have been most severely impacted by the novel coronavirus (COVID-19) pandemic. This project aims to assess the impact of patient navigation as an intervention tool in patient populations that are most at risk for delayed follow-up. The investigators hypothesize that patient navigation services may be an effective way to mitigate the impact of the pandemic by decreasing the risk of a delayed breast cancer diagnosis and promoting timely diagnostic follow-up.

DETAILED DESCRIPTION:
Patients who meet the study selection criteria will be randomized into two groups in a 1:1 ratio: the usual care group and the intervention group. Initially, patients will be invited to participate in the study via a brief statement included in the patient result letter informing patients of their abnormal screening mammogram result. The patient navigator will then follow up with each patient who expresses interest in the study via telephone to reiterate the details of the project, answer any questions that the patients might have, and invite the patients to participate in the project if the patients meet the study inclusion criteria. Informed consent will be obtained from the study participants.

The primary role of the patient navigator will be to identify and address barriers to accessing timely diagnostic care. The patient navigator's duties will also include providing an array of services aimed at improving health care access and engagement, including appointment reminder phone calls, health education, assistance with scheduling appointments, providing information about available transportation options to the clinic sites (e.g., shuttle service provided by the institution), helping patients to connect with language interpretation services, providing assistance with resolving insurance issues, and motivating and coaching patients on the importance of timely follow-up of abnormal breast imaging results. The services provided by the patient navigator will be tailored to the specific needs of each patient and will be aimed at helping patients to overcome personal, cultural and systemic barriers to successfully completing follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have an abnormal screening mammogram (i.e. given a Breast Imaging-Reporting and Data System [BI-RADS] assessment category of 0) at the investigators' institution during the study period and have not yet undergone diagnostic evaluation

Exclusion Criteria:

* Any study participant who is unable to provide consent to participate in the study will be excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2022-07-18 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Diagnostic follow-up rates | 30 days after the screening mammogram
  The follow-up rates for patients with an abnormal screening mammogram will be calculated. This will be expressed as the percentage of patients who follow-up within 30 days after the abnormal screening mammogram.

SECONDARY OUTCOMES:
Anxiety level as assessed by the Spielberger State-Trait Anxiety Inventory | 1 day prior to the scheduled diagnostic appointment
  The study participants' anxiety level will be assessed using the 6-item short form of the state scale of the Spielberger State-Trait Anxiety Inventory (STAI).
Breast cancer worry as assessed by the Lerman Breast Cancer Worry Scale | 1 day prior to the scheduled diagnostic appointment
  The study participants' level of worry about breast cancer will be assessed using the 3-item Lerman Breast Cancer Worry Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Eniola Oluyemi, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Breast Imaging clinics, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No